CLINICAL TRIAL: NCT00310882
Title: Involvement of Endogenous Digitalis-like Compounds in Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Tanir Allweiss, Hadassah Medical Organization
Other Study IDs: 297-31.3-06-HMO-CTIL
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-05

CONDITIONS: Breast Neoplasms; Fibrocystic Disease of Breast; Mammaplasty
Keywords: breast cancer; digitalis like compounds; prognostic factor
MeSH Terms: conditions — Breast Neoplasms; Fibrocystic Breast Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The endogenous digitalis-like compounds (DLC)are steroid hormones synthesized and released from the adrenal gland.They are integrated in the feed-back system of the Hypothalami-Pituitary-Adrenal gland axis.One of their remarkable function is to induce apoptosis in malignant cells. Recently, accumulating data point to the possibility of using synthetic DLC as new anti-cancer drugs. Less is known about the endogenous metabolism of these compounds in cancer patients.

Proceeding from preliminary clinical data which demonstrated significantly reduced DLC plasma levels in breast cancer patients and from in vitro data which showed an impaired release of DLC towards stress stimuli in athymic nude mice,we put up the hypothesis that a latent adrenal insufficiency with low DLC levels facilitates the induction and progression of tumor diseases.

DETAILED DESCRIPTION:
To pursue this question about endogenous DLC metabolism in cancer patients we intend to start with the measurement of DLC plasma levels in breast cancer patients at the time of first diagnosis and compare them to women with benign breast disease as well as healthy women.

Aim of the Study

* To evaluate the basal DLC plasma concentrations in cancer patients at the time of first diagnosis and the function of the HPA axis, with focussing on breast cancer patients.
* To analyze a potential change of HPA function and, in parallel, DLC plasma concentrations in the course of therapy, with special respect to treatment failure.
* To establish a potential correlation between DLC plasma concentrations and risk factors in BC.

Patients and Methods

Patients:

I. 50 - (100) patients with breast cancer at the time of first diagnosis

II. 50 - (100) patients with a benign disease of the breast

III. 50 - (100) women undergoing plastic surgery of the breast

IV. 50 - (100) women who need no further exploration after visit in ambulance (=normal population)

V. additionally a group of 25 - 50 students (age 20-40) will be analyzed in a pilot study

Methods:

Time-schedule for Group I (Group II. - IV. alike, according to disease and/or situation)

* Day of first presentation of the woman at the clinic
* Day of first diagnosis, i.e. biopsy/FNA
* Day of start of treatment: operation, chemo-/radiotherapy (tst = 0)
* Day + 30, + 60, + 90
* 6 month and 1 year after start of treatment

The Group V. (students) will be analyzed in a special schedule, preceding the study 1-2 months:

* 4 weeks before an important exam
* a day before the exam (-3 days)
* a day after the exam (+ 3 days)
* 2 weeks after the exam
* 6 weeks after the exam

Parameters

Biochemistry (Group I. - V.)

* Basal DLC plasma concentration
* Basal serum Cortisol concentration
* Basal plasma ATCH concentration
* Basal Aldosterone/Renin concentration
* Electrolytes (potassium, sodium, calcium, chloride)

Pathology/Immunohistochemistry (Group I. + II., when benign, including last 4 points)

* Tumor size
* lymph node status
* E/P receptors
* Grade
* HER2/neu
* Bcl-2
* Ki67
* p53

Radiology (Group I.)

If abdominal CT available measurement of size of the adrenal glands

Endocrinologic tests (Group I. - IV.)

* Dexamethasone-test (low dose):

  * 2 mg Dexamethasone p.o. at 24:00
  * measurement of Cortisol and DLC at 8:00 the next morning
* ACTH-test:

  * basal plasma concentrations of Cortisol, DLC and ACTH
  * administration of 250 µg ACTH (Synachten®) i.v.
  * measurement of Cortisol and DLC after 30 min. and 60 min.
* Facultative: Metapyrone test

at following time intervals:

1. Dexamethasone-test

   * around the time of first presentation (± 5 days)
   * around the time of start of treatment (± 5 days); corresponding times for Group II.- IV.
   * Day + 30, +60, +90
   * 6 month and a year after start of treatment
2. ACTH-test

   * On the day of first presentation
   * On the day of start of treatment; corresponding times for Group II.- IV.
   * Day + 30, +60, +90
   * 6 months and one year after start of treatment

Psychometric test for Stress Evaluation (Group I. - V.)

* at the day of first presentation (Students: in between the last 2 weeks before an exam)
* at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* first visit to a Breast Disease Ambulance for consultation
* no pregnancy

Exclusion Criteria:

* no severe heart disease (EF > 40%)
* no therapy with digitalis
* no acute/chronic inflammatory disease (e.g. RA, M. Crohn)
* no dysfunction of the Hypothalamo-Pituitary-Adrenal system
* no severe mental disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with first diagnosis of Breast Cancer or a benign Breast Disease
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2006-05; Study Completion 2008-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Heidrun Weideman, Principal Investigator — Hadassah Hebrew University Medical Centers
Locations (1):
- Hadassah Hebrew University Medical Centers, Jerusalem, Israel